CLINICAL TRIAL: NCT01158404
Title: Phase 1 Study of a Notch Inhibitor in Patients With Advanced Cancer
Brief Title: Notch Inhibitor in Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13284; I3F-MC-JSRB (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-06

CONDITIONS: Advanced Cancer
Keywords: Metastatic Cancer; Solid Tumors
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY900009 (Experimental): Dose escalation phase: 2 milligrams (mg), 4 mg, 8 mg, 15 mg, 30 mg, 45 mg and 60mg LY900009 administered orally 3 times per week (Monday, Wednesday, Friday) for 4 weeks of a 28-day cycle.
  Dose confirmation phase: 30 mg LY900009 administered orally 3 times per week (Monday, Wednesday, Friday) for 4 weeks of a 28-day cycle.
  Participants experiencing clinical benefit may continue treatment unless discontinuation criteria are met.
  Interventions: Drug: LY900009 - Dose Escalation Phase (Part A); Drug: LY900009 - Dose Confirmation Phase (Part B)

INTERVENTIONS:
Drug: LY900009 - Dose Escalation Phase (Part A) — 2 milligrams (mg), 4 mg, 8 mg, 15 mg, 30 mg, 45 mg and 60mg LY900009 administered orally 3 times per week (Monday, Wednesday, Friday) for 4 weeks of a 28-day cycle.
  Participants experiencing clinical benefit may continue treatment unless discontinuation criteria are met.
  Other Names: Notch Inhibitor
Drug: LY900009 - Dose Confirmation Phase (Part B) — 30 mg LY900009 orally 3 times per week (Monday, Wednesday, Friday) for 4 weeks of a 28-day cycle.
  Participants experiencing clinical benefit may continue treatment unless discontinuation criteria are met.
  Other Names: Notch Inhibitor

SUMMARY:
The objective of this phase 1 study is to evaluate the safety and tolerability of Notch Inhibitor in participants with advanced cancer. This study includes dose escalation and dose confirmation components.

ELIGIBILITY:
Inclusion Criteria:

* The participants must be, in the judgment of the investigator, an appropriate candidate for experimental therapy after available standard therapies have ceased to provide clinical benefit for their disease.
* The participants must have histological or cytological evidence of cancer, either a solid tumor or a lymphoma, which is advanced and/or metastatic.
* Have adequate organ function including:

  * Hematologic: Absolute neutrophil count (ANC) ≥1.5 x 10⁹/liter (L), platelets ≥100 x 10⁹/L, and hemoglobin ≥8 grams/deciliter (g/dL).
  * Hepatic: Bilirubin ≤1.5 times upper limits of normal (ULN) and alanine aminotransferase (ALT) ≤3.0 times ULN.
  * Renal: Serum creatinine ≤1.5 times ULN.
* Have a performance status less than or equal to 1 for Dose Escalation and less than or equal to 2 for Dose Confirmation on the Eastern Cooperative Oncology Group (ECOG) scale.
* Have discontinued all previous therapies for cancer (including chemotherapy, radiotherapy, immunotherapy, and investigational therapy) for at least 21 days for myelosuppressive agents or 14 days for nonmyelosuppressive agents prior to receiving study drug, and recovered from the acute effects of therapy (treatment-related toxicity resolved to baseline) except for residual alopecia.
* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the trial and for 3 months following the last dose of study drug.
* Females with childbearing potential must have a negative serum pregnancy test within 7 days of the first dose of study drug.

Exclusion Criteria:

* Have received treatment with a drug that has not received regulatory approval for any indication within 14 or 21 days of the initial dose of study drug for a nonmyelosuppressive or myelosuppressive agent, respectively.
* Have serious preexisting medical conditions that, in the judgment of the investigator, would preclude participation in this study (for example, inflammatory bowel disease or history of major surgical resection involving the stomach or small bowel).
* Have malabsorptive syndromes, enteropathies, gastroenteritis (acute or chronic), or diarrhea (acute or chronic).
* Females who are pregnant or lactating.
* Have Central Nervous System (CNS) malignancy or metastasis.
* Have an acute leukemia.
* Have active bacterial, fungal and/or known viral infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT -5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee

REFERENCES:
- [Derived] Pant S, Jones SF, Kurkjian CD, Infante JR, Moore KN, Burris HA, McMeekin DS, Benhadji KA, Patel BKR, Frenzel MJ, Kursar JD, Zamek-Gliszczynski MJ, Yuen ESM, Chan EM, Bendell JC. A first-in-human phase I study of the oral Notch inhibitor, LY900009, in patients with advanced cancer. Eur J Cancer. 2016 Mar;56:1-9. doi: 10.1016/j.ejca.2015.11.021. Epub 2016 Jan 19. PMID 26798966

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Any participant who completed Cycle 1 or discontinued due to an adverse event (AE) in Part A is considered a completer. Any participant who completed cycle 1 or discontinued due to an AE or progressive disease in Part B was considered a completer.
Groups:
- 2 mg LY900009 - Dose Escalation Phase (Part A): 2 milligram (mg) LY900009 administered orally 3 times per week (every Monday, Wednesday, and Friday) for 4 weeks of a 28-day cycle.
- 4 mg LY900009 - Dose Escalation Phase (Part A): 4 mg LY900009 administered orally 3 times per week (every Monday, Wednesday, and Friday) for 4 weeks of a 28-day cycle.
- 8 mg LY900009 - Dose Escalation Phase (Part A): 8 mg LY900009 administered orally 3 times per week (every Monday, Wednesday, and Friday) for 4 weeks of a 28-day cycle.
- 15 mg LY900009 - Dose Escalation Phase (Part A): 15 mg LY900009 administered orally 3 times per week (every Monday, Wednesday, and Friday) for 4 weeks of a 28-day cycle.
- 30 mg LY900009 - Dose Escalation Phase (Part A); 30 mg LY900009 - Dose Confirmation Phase (Part B): 30 mg LY900009 administered orally 3 times per week (every Monday, Wednesday, and Friday) for 4 weeks of a 28-day cycle.
- 45 mg LY900009 - Dose Escalation Phase (Part A): 45 mg LY900009 administered orally 3 times per week (every Monday, Wednesday, and Friday) for 4 weeks of a 28-day cycle.
- 60 mg LY900009 - Dose Escalation Phase (Part A): 60 mg LY900009 administered orally 3 times per week (every Monday, Wednesday, and Friday) for 4 weeks of a 28-day cycle.
Period: Overall Study
Arm/Group | 2 mg LY900009 - Dose Escalation Phase (Part A) | 4 mg LY900009 - Dose Escalation Phase (Part A) | 8 mg LY900009 - Dose Escalation Phase (Part A) | 15 mg LY900009 - Dose Escalation Phase (Part A) | 30 mg LY900009 - Dose Escalation Phase (Part A) | 45 mg LY900009 - Dose Escalation Phase (Part A) | 60 mg LY900009 - Dose Escalation Phase (Part A) | 30 mg LY900009 - Dose Confirmation Phase (Part B)
Started | 3 | 4 | 3 | 3 | 6 | 5 | 3 | 8
Received at Least 1 Dose of Study Drug | 3 | 4 | 3 | 3 | 6 | 5 | 3 | 8
Completed | 3 | 3 | 3 | 3 | 3 | 4 | 2 | 6
Not Completed | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- 2 mg LY900009 - Dose Escalation Phase (Part A): 2 mg LY900009 administered orally 3 times per week (every Monday, Wednesday, and Friday) for 4 weeks of a 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | 2 mg LY900009 - Dose Escalation Phase (Part A) | 4 mg LY900009 - Dose Escalation Phase (Part A) | 8 mg LY900009 - Dose Escalation Phase (Part A) | 15 mg LY900009 - Dose Escalation Phase (Part A) | 30 mg LY900009 - Dose Escalation Phase (Part A) | 45 mg LY900009 - Dose Escalation Phase (Part A) | 60 mg LY900009 - Dose Escalation Phase (Part A) | 30 mg LY900009 - Dose Confirmation Phase (Part B) | Total
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 6 | 5 | 3 | 8 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (5.5) | 54.0 (9.0) | 66.0 (14.2) | 57.3 (13.6) | 62.5 (8.6) | 58.4 (21.9) | 55.7 (13.7) | 57.5 (9.8) | 58.8 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 3 | 3 | 4 | 1 | 2 | 8 | 27
  Male | 1 | 0 | 0 | 0 | 2 | 4 | 1 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 4 | 3 | 3 | 6 | 5 | 3 | 7 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  White | 2 | 4 | 3 | 2 | 6 | 5 | 3 | 7 | 32
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 4 | 3 | 3 | 6 | 5 | 3 | 8 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Effects
Description: Clinically significant effects are study drug related serious adverse events (SAEs) and study drug related treatment emergent adverse events (TEAEs). A summary of all SAEs and all other non-SAEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline to study completion up to 18.7 weeks
Population: All enrolled participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 60 mg LY900009 - Part A: Dose Escalation: 60 mg LY900009 administered orally 3 times per week (every Monday, Wednesday, and Friday) for 4 weeks of a 28-day cycle.
Arm/Group | 2 mg LY900009 - Dose Escalation Phase (Part A) | 4 mg LY900009 - Dose Escalation Phase (Part A) | 8 mg LY900009 - Dose Escalation Phase (Part A) | 15 mg LY900009 - Dose Escalation Phase (Part A) | 30 mg LY900009 - Dose Escalation Phase (Part A) | 45 mg LY900009 - Dose Escalation Phase (Part A) | 60 mg LY900009 - Part A: Dose Escalation | 30 mg LY900009 - Dose Confirmation Phase (Part B)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 6 | 5 | 3 | 8
Participants
  SAEs | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  TEAEs | 2 | 1 | 3 | 3 | 5 | 5 | 2 | 6

2. Secondary Outcome: Recommended Dose Range for Phase 2 Studies
Description: Recommended Phase 2 dose was determined by the maximum tolerated dose (MTD). MTD is the highest dose with <33% of participants having a dose-limiting toxicity (DLT) during Cycle 1. DLT is an adverse event (AE) occurring for a participant enrolled in Part A that is likely related to the study drug and fulfills any 1 of the following: Common Terminology Criteria for AE (CTCAE, Version 4.02) Grade 3 or 4 nonhematologic toxicity except for Grade 3 nausea, vomiting or electrolyte disturbance; Grade 3 nausea, vomiting or electrolyte disturbance that persists more than 2 days despite maximal supportive intervention; Grade 4 hematological toxicity that persists more than 5 days; Grade 3 or 4 thrombocytopenia with bleeding; Grade 3 or 4 neutropenia with fever. A DLT can be declared if a participant experiences increasing toxicity during treatment.
Time Frame: Predose up to 28 days in Cycle 1
Population: All enrolled participants who received at least one dose of study drug during dose escalation phase.
Measure: Number; unit: milligrams (mg)
Groups:
- LY900009 - Dose Escalation Phase (Part A): 2 mg, 4 mg, 8 mg, 15mg, 30 mg, 45 mg and 60 mg LY900009 administered orally 3 times per week (every Monday, Wednesday, and Friday) for 4 weeks of a 28-day cycle.
Arm/Group | LY900009 - Dose Escalation Phase (Part A)
Number analyzed (Participants) | 27
milligrams (mg) | 30

3. Secondary Outcome: Percentage of Participants With a Best Overall Response of Stable Disease or Better (Document the Antitumor Activity)
Description: Best overall response of stable disease or better is complete response (CR) + partial response (PR) + stable disease (SD) as classified by the investigator according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines (version 1.1). CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. Percentage of Participants with a best overall response of SD or better is calculated as a total number of participants with CR or PR or SD divided by the total number of participants treated then multiplied by 100.
Time Frame: Baseline to measured progressive disease up to 15.1 weeks
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 2 mg LY900009 - Dose Escalation Phase (Part A) | 4 mg LY900009 - Dose Escalation Phase (Part A) | 8 mg LY900009 - Dose Escalation Phase (Part A) | 15 mg LY900009 - Dose Escalation Phase (Part A) | 30 mg LY900009 - Dose Escalation Phase (Part A) | 45 mg LY900009 - Dose Escalation Phase (Part A) | 60 mg LY900009 - Dose Escalation Phase (Part A) | 30 mg LY900009 - Dose Confirmation Phase (Part B)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 6 | 5 | 3 | 8
percentage of participants | 33.3 | 0 | 66.7 | 33.3 | 16.7 | 0 | 0 | 0

4. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-time Curve of LY900009 From Time Zero to Infinity [AUC(0-infinity)]
Description: The geometric mean AUC(0-infinity) for each dose group is reported following a single dose of LY900009.
Time Frame: Day1: Pre-dose, 0.5 hours (hr), 1 hr, 3-4 hr, 6-8 hr and 24-30 hours post-dose
Population: All enrolled participants who received the study drug and had sufficient pharmacokinetic (PK) data to calculate AUC(0-infinity).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliters (ng*h/mL)
Groups:
- 30 mg LY900009 - Dose Escalation/Confirmation Phase (Part A,B): 30 mg LY900009 administered orally 3 times per week (every Monday, Wednesday, and Friday) for 4 weeks of a 28-day cycle.
Arm/Group | 2 mg LY900009 - Dose Escalation Phase (Part A) | 4 mg LY900009 - Dose Escalation Phase (Part A) | 8 mg LY900009 - Dose Escalation Phase (Part A) | 15 mg LY900009 - Dose Escalation Phase (Part A) | 30 mg LY900009 - Dose Escalation/Confirmation Phase (Part A,B) | 45 mg LY900009 - Dose Escalation Phase (Part A) | 60 mg LY900009 - Dose Escalation Phase (Part A)
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 14 | 5 | 3
nanograms*hour/milliliters (ng*h/mL) | NA (NA) — For n=2, range (8.37 - 35.6) was reported. | 31.6 (48) | 76.2 (123) | 121 (59) | 315 (71) | 547 (32) | 1240 (53)

5. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY900009
Description: The geometric mean Cmax for each dose group is reported following a single dose of LY900009.
Time Frame: Day1: Pre-dose, 0.5 hours (hr), 1 hr, 3-4 hr, 6-8 hr and 24-30 hours post-dose
Population: All enrolled participants who received the study drug and had sufficient pharmacokinetic (PK) data to calculate Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | 2 mg LY900009 - Dose Escalation Phase (Part A) | 4 mg LY900009 - Dose Escalation Phase (Part A) | 8 mg LY900009 - Dose Escalation Phase (Part A) | 15 mg LY900009 - Dose Escalation Phase (Part A) | 30 mg LY900009 - Dose Escalation/Confirmation Phase (Part A,B) | 45 mg LY900009 - Dose Escalation Phase (Part A) | 60 mg LY900009 - Dose Escalation Phase (Part A)
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 14 | 5 | 3
nanograms/milliliter (ng/mL) | 4.03 (122) | 11.7 (70) | 20.2 (68) | 27.4 (50) | 71.2 (104) | 96.2 (37) | 158 (35)

ADVERSE EVENTS:
Time Frame: Up To 18.7 Weeks
Description: All enrolled participants who received at least one dose of study drug.
Arm/Group | 2 mg LY900009 - Dose Escalation Phase (Part A) | 4 mg LY900009 - Dose Escalation Phase (Part A) | 8 mg LY900009 - Dose Escalation Phase (Part A) | 15 mg LY900009 - Dose Escalation Phase (Part A) | 30 mg LY900009 - Dose Escalation/Confirmation Phase (Part A,B) | 45 mg LY900009 - Dose Escalation Phase (Part A) | 60 mg LY900009 - Dose Escalation Phase (Part A)
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/4 | 0/3 | 1/3 | 7/14 | 3/5 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/4 | 3/3 | 3/3 | 14/14 | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg LY900009 - Dose Escalation Phase (Part A) (N=3) | 4 mg LY900009 - Dose Escalation Phase (Part A) (N=4) | 8 mg LY900009 - Dose Escalation Phase (Part A) (N=3) | 15 mg LY900009 - Dose Escalation Phase (Part A) (N=3) | 30 mg LY900009 - Dose Escalation/Confirmation Phase (Part A,B) (N=14) | 45 mg LY900009 - Dose Escalation Phase (Part A) (N=5) | 60 mg LY900009 - Dose Escalation Phase (Part A) (N=3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg LY900009 - Dose Escalation Phase (Part A) (N=3) | 4 mg LY900009 - Dose Escalation Phase (Part A) (N=4) | 8 mg LY900009 - Dose Escalation Phase (Part A) (N=3) | 15 mg LY900009 - Dose Escalation Phase (Part A) (N=3) | 30 mg LY900009 - Dose Escalation/Confirmation Phase (Part A,B) (N=14) | 45 mg LY900009 - Dose Escalation Phase (Part A) (N=5) | 60 mg LY900009 - Dose Escalation Phase (Part A) (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 9 (9) | 3 (4) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 6 (7) | 2 (2) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 2 (2) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 1 (2) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyposmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days